CLINICAL TRIAL: NCT02175264
Title: Genetic Basis of Non Syndromic Congenital Diaphragmatic Hernia
Acronym: HCD GENE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: CRC12074
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Isolated Non Syndromic Left CDH With Postero Lateral Diaphragmatic Defect With Good Perinatal Outcome
Keywords: Isolated non syndromic CDH
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients and Families with isolated non syndromic CDH cases
  Interventions: Genetic: Blood sample

INTERVENTIONS:
Genetic: Blood sample

SUMMARY:
In isolated congenital diaphragmatic hernia (CDH), recurrent risk is low suggesting the occurrence of novo mutations (dominant or recessive). Our objective is to test this hypothesis by combining the search for pathogenic genomic alteration and intragenic mutations through whole exome sequencing in a homogenous group of patients.

DETAILED DESCRIPTION:
To elucidate the genetic basis of non syndromic congenital diaphragmatic hernia in a sub group of individuals with similar phenotype: Isolated CDH presenting with postero-lateral-left diaphragmatic defect with good perinatal outcome (n=16) To establish the prevalence of the identified gene(s) in a cohort of identical patients (n=30)

Two complementary approaches will be used:

* Search for pathogenic genomic alterations using microarrays (~2.106 markers (SNP and CNV) in 16 trios (affected child and 2 parents).
* Sequencing of the whole exome from patient genomic DNA (n=16)
* Selection of unknown or very rare variants according to different criteria: recessive or dominant model, prediction of their pathogenicity, filtered on genes already known in CDH or involved in diaphragmatic development and non annotated CNV or variants of new gene(s) shared by different patients.
* Variants will be validated by Sanger sequencing (for intragenic variants) or quantitative PCR (for CNV) on CDH cases and their parents as well as their absence on 100 controls.

ELIGIBILITY:
Inclusion Criteria:

* Families with one (or more) non syndromic CDH child
* Signed consent form

Exclusion Criteria:

* Syndromic CDH or associated with a known karyotype anomaly
* No signed consent form
* Not affiliated to French social security

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Babies with CDH who delivered if centers included in the "Centre For Rare Disease for Congenital Diaphragmatic Hernia"
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
genes responsible for isolated CDH | One year

SECONDARY OUTCOMES:
prevalence of new identified genes in a cohort of CDH | One year

CONTACTS AND LOCATIONS:
Overall Officials: Judith Melki, MD-PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hopital béclère, Clamart, France